CLINICAL TRIAL: NCT06899308
Title: Health Surveillance at Constructor University Bremen (CUB) to Assess Students' and HAW-Hamburg Employees' Health and Wellbeing - Explanatory Sequential Mixed-Methods Approach
Brief Title: Health Surveillance at Constructor University Bremen (CUB) and Among HAW-Hamburg Employees
Acronym: CUB-HS2025
Status: Recruiting | Type: Observational
Sponsor: Jacobs University Bremen gGmbH (Other)
Collaborators: Hamburg University of Applied Sciences/Hochschule für Angewandte Wissenschaften Hamburg (HAW Hamburg) (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Sonia Lippke, Professor of Health Promotion and Prevention, Jacobs University Bremen gGmbH
Other Study IDs: CUB2025-03-12
Record Dates: First submitted 2025-03-11; First posted 2025-03-27 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Social Isolation or Loneliness; Anxiety; Anxiety Depression (Mild or Not Persistent); Health Behavior; Observational Study; Stress, Psychological; Emotional Stress; Life Stress; Psychological Stress; Stress, Emotional; Stress (Psychology); Substance Abuse; Substance Addiction; Substance Dependence; Substance Use
Keywords: Healthy students; Health literacy; Disability; Age; Gender; Study characteristics; PHQ-4; Self-efficacy; Satisfaction with Life Scale (SWLS); Subjective health status; Student satisfaction; UCLA-LS; HEI-Stress; Mixed Method
MeSH Terms: conditions — Social Isolation; Anxiety Disorders; Lymphoma, Follicular; Health Behavior; Stress, Psychological; Substance-Related Disorders; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- students: Students at Constructor University Bremen

SUMMARY:
The aim of Health Surveillance is to analyze and describe the state of health of students at Constructor University, key influencing factors and individual resources by using mixed-method design.

DETAILED DESCRIPTION:
The aim of Health Surveillance plus the additional research by means of qualitative interviews is to analyze and describe the state of stress and health of students at Constructor University (CU) by using a mixed-methods approach, as well as explore the association and mechanism between stress and health of students at CU (and employees at HAW Hamburg), key influencing factors and individual resources. In areas where there is a need for action, the Health Surveillance plus this project the additional qualitative interviews can provide detailed insights and/or in-depth analyses. The Health Surveillance thus provides information on health-related topics and delivers scientifically sound information as a basis for health-promoting discussions in the subsequent follow-up process at various levels (e.g. faculties and departments). In addition, the Health Surveillance plus the additional interviews at CU contributes to comparability with surveys at other German universities through the use of validated and standardized measuring instruments and in-depth qualitative interviews with qualitative content analysis.

Main hypotheses are

1. The Health Surveillance gives insights into state of stress and health of students at CU, key influencing factors and individual resources by using a mixed-methods approach.
2. With the Health Surveillance the health-promotion at CU by using a mixed-methods approach, as well as explore the association and mechanism between stress and health of students at CU (and employees at HAW Hamburg), can be guided and promotion of mental health (including the reduction of loneliness and discrimination) can be strengthened.
3. The health of students (and employees at HAW Hamburg), their perceived stress, loneliness and discrimination/minorization (disadvantage) as well as substance use interrelates with participation in health promoting activities?
4. Recommendations can be derived for qualification and skills training of multipliers for health-promoting behavior (e.g., J-peers)?

ELIGIBILITY:
Inclusion Criteria:

* English language skills
* Reading and writing skills
* Internet access
* Student status
* Consent to participate in the study

Exclusion Criteria:

* Illiteracy
* Massively limited cognitive abilities ( i.e. linguistic components of the digital offerings must be able to be used, and questionnaires completed, or interviews participated in) and severe psychiatric disorders (e.g., severe depression)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This project contains two phases, the first one is quantitative phase (finished) and the second one is qualitative phase (Dec 2025-Dec 2026). All Constructor University students and employees at HAW Hamburg who wish to take part in the study will be included. In the quantitative phase, Iinclusion criteria are englsih English language for CU students and German language for HAW employees, reading and writing skills, internet access and student status. In the qualitative phase, the inclusion criteria are English or Chinese language and between 18-30 years old. Before the start of the survey period and directly before the start of the online survey or interview, all participants will receive all relevant study information and actively declare their consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 363 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Loneliness | Baseline
  University of California Los Angelese Loneliness Scale (UCLA-LS) - 3 Items (Schobin, Arriagada & Gibson-Kunze, 2024), Range 1 (never/nie) - 5 (very often/sehr oft), higher scores mean a worse outcome
  Loneliness in private and study context - 9 Items (Techniker Krankenkasse, 2024), Range 1 (often) - 4 (never), higher scores mean better outcomes
Health literacy | Baseline
  Health literacy - 10 Items (Lenartz, Söllner & Rudinger, 2014), Range 1 (does not apply/trifft überhaupt nicht zu) - 4 (does fully apply/trifft genau zu), higher scores mean a better outcome

SECONDARY OUTCOMES:
Depression and anxiety | Baseline
  Patient Health Questionnaire (PHQ-4) - 4 Items (Kroenke, Spitzer, Williams & Löwe, 2009), Range 0 (not at all/überhaupt nicht) - 3 (nearly every day/beinahe jeden Tag), higher scores mean worse outcome
Subjective health status | Baseline
  Subjective health status- 1 Item (WHO, 1996); Range 1 (very good/sehr gut) - 5 (very poor/schlecht), higher score means worse outcome
Student satisfaction | Baseline
  Student satisfaction - 1 Item (Westermann, Heise, Spies & Trautwein, 1996), Range 0 (not at all satisfied/gar nicht zufrieden) - 100 (completely satisfied/vollkommen zufrieden), higher scores mean better outcome
HEI-Stress | Baseline
  Higher Education Institution Stress (HEI-Stress) - 3 Items (Schmidt, Sieverding, Scheiter & Obergfell, 2013), Range 0 (not at all stressed/gar nicht gestresst) - 100 (very stressed/sehr gestresst), higher scores mean worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Lippke, PhD, Principal Investigator — Constructor University Bremen gGmbH & Bremen International Graduate School of Social Sciences, Germany
Locations (2):
- Germany (2):
  - Constructor University (formerly known as Jacobs University), Bremen
  - Constructor University Bremen, Bremen

IPD SHARING:
Plan to Share IPD: No
due to data security

REFERENCES:
- See also: World Health Organization (WHO) (Hrsg.). (2996). Health interview survey: Towards international harmonization of methods and instruments. World Health Organization, Regional Office for Europe, Kopenhagen. — https://iris.who.int/bitstream/handle/10665/107328/9789289013222-eng.pdf?sequence=1&isAllowed=y
- See also: Burian, J., Lehnchen, J. Deptolla, Z., Heinrichs, K., Stock, C. (2023). Abschlussbericht zum Vorhaben "Studienbedingungen und (psychische) Gesundheit Studierender: Weiterentwicklung und Erprobung des Bielefelder Fragebogens zu Studienbedingungen — https://www.dguv.de/projektdatenbank/0460/fp460_fin_abschlussbericht_mu.pdf
- See also: Kroenke, K., Spitzer, R. L., Williams, J. B. W., & Löwe, B. (2009). An Ultra-Brief Screening Scale for Anxiety and Depression: The PHQ-4. Psychosomatics, 50(6), 613-621. DOI: — https://www.researchgate.net/publication/40483064_An_Ultra-Brief_Screening_Scale_for_Anxiety_and_Depression_The_PHQ-4
- See also: Schobin, J, Arriagada, C., Gibson-Kunze, M. (2024). Einsamkeitsbarometer 2024. Langzeitentwicklund von Einsamkeit in Deutschland. Einsamkeitsbarometer 2024, 1, 1-78. Bundesministerium für Familie, Senioren, Frauen und Jugend (BMFSFJ) (Hrsg.). — https://www.bmfsfj.de/resource/blob/240528/5a00706c4e1d60528b4fed062e9debcc/einsamkeitsbarometer-2024-data.pdf
- See also: Techniker Krankenkasse. (2024). Einsamkeitsreport 2024. Techniker Krankenkasse: Hamburg (Hrsg.). — https://www.tk.de/resource/blob/2186830/73239d0d1b389491c47f1bf7960ed254/2024-tk-einsamkeitsreport-data.pdf
- See also: SOEP-IS Group (2022). SOEP-IS 2020 - Fragebogen für die SOEP-Innovations-Stichprobe. SOEP Survey Papers 1143: Series A - Survey Instruments (Erhebungsinstrumente). Berlin: DIW Berlin/SOEP. — https://www.diw.de/documents/publikationen/73/diw_01.c.844972.de/diw_ssp1143.pdf
- See also: Deutsches Zentrum für Hochschul- und Wissenschaftsforschung GmbH (DZHW) (2021). Die Studierendenbefragung in Deutschland. Grundprogramm Modul A. Hannover: FDZ-DZHW. — https://doi.org/10.21249/DZHW:sid2021-ins1-att1:1.0.0
- See also: Janke, S. & Glöckner-Rist, A. (2014). Deutsche Version der Satisfaction with Life Scale (SWLS). Zusammenstellung sozialwissenschaftlicher Items und Skalen (ZIS) — https://zis.gesis.org/skala/Janke-Gl%C3%B6ckner-Rist-Deutsche-Version-der-Satisfaction-with-Life-Scale-%28SWLS%29
- See also: Knispel, J., Wittneben, L., Slavchova, V., & Arling, V. (2021). Skala zur Messung der berufli-chen Selbstwirksamkeitserwartung (BSW-5-Rev). Zusammenstellung sozialwissenschaftlicher Items und Skalen (ZIS). — https://doi.org/10.6102/ZIS303